CLINICAL TRIAL: NCT06864156
Title: Evaluation of MicroRNAs and Vitamin B12 Expression in Subjects with Neurologic Symptoms of Depression, Anxiety and Fatigue in Long COVID-19
Status: Recruiting | Type: Observational
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, Alfonso B. Alfaro, Principal Investigator, Instituto Nacional de Rehabilitacion
Other Study IDs: 03/24 AD 2025
Record Dates: First submitted 2025-02-26; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Long COVID; Long COVID Syndrome
Keywords: anxiety; depression; fatigue; microRNAs; vitamin b12; long covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Anxiety Disorders; Depression; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Long COVID: With presence of neurological symptoms of depression, anxiety and fatigue associated with COVID-19 three months after the first day with symptoms of acute infection
- Control: Not presented symptoms associated with COVID-19 twelve weeks after the first day with symptoms of acute infection

SUMMARY:
At the moment, the number of people with long COVID is unkown because there is still no effective diagnosis. This is why is very important to analyze the most common symptoms, which are: depression, anxiety and fatigue. This project seeks to analyze some blood components of people with long COVID, such as microRNAs and vitamin B12, in order to identify the body processes that changed after COVID-19 and thereby design better therapies and diagnostic methods focused on each of them.

The hypothesis is that the expression of miR-21, -146a and -155 will be overexpressed as well as there will be a deficiency of vitamin B12 in serum in subjects suffering from long COVID with neurological symptoms of depression, anxiety and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with confirmed diagnosis of COVID-19 by SARS-CoV-2 infection by PCR or antigen testing.
* With presence of neurological symptoms of depression, anxiety and fatigue associated with COVID-19 after three months from the first day of acute infection symptoms.

Exclusion Criteria:

* Subjects who have presented symptoms of acute infection in the last twelve weeks.
* Subjects who present diagnostic premorbid neurological alterations.
* Subjects who do not have at least 2 doses of COVID-19 vaccine, with last application date equal or older than 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with symptoms of depression, anxiety and fatigue after having had COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change of microRNA expression between long COVID group and control group | immediately after the blood extraction
Change of vitamin B12 concentration between long COVID group and control group | immediately after the blood extraction
Link the expression of microRNAs with the score obtained in the instruments to evaluate depression, anxiety and fatigue | immediately after the blood extraction
Link the concentration of vitamin B23 with the score obtained in the instruments to evaluate depression, anxiety and fatigue. | immediately after the blood extraction

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Rehabilitación, Mexico City, Mexico City, Mexico